CLINICAL TRIAL: NCT02515877
Title: Modulation of the Expression of Papillomavirus (HPV) Oncoproteins to Major the Radiosensitivity: Phase I Trial Combining an Antiviral Agent VISTIDE and Radiochemotherapy in Cervical Cancers
Brief Title: Modulation of the Expression of Papillomavirus (HPV) Oncoproteins to Major the Radiosensitivity: Trial Combining an Antiviral Agent VISTIDE and Radiochemotherapy in Cervical Cancers
Acronym: HPV-RX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-005505-21; 2007/1297 (Other: CSET number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Brachytherapy; Cidofovir; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy + Vistide + Chemoterapy (Experimental)
  Interventions: Radiation: External radiotherapy + curietherapy; Drug: Vistide; Drug: Carboplatin

INTERVENTIONS:
Radiation: External radiotherapy + curietherapy — External radiotherapy: 45 Gy in 5 weeks Curietherapy: 15Gy
Drug: Vistide — VISTIDE® (mg/kg) Level 1: 1mg/kg Level 2: 2,5 mg/kg Level 3: 5 mg/kg Level 4: 6,5 mg/kg
Drug: Carboplatin — AUC= 2,5 (Calvert formula)

SUMMARY:
The treatment of cervical tumors depends on the stage of the disease. In advanced forms (nodal and / or local extension to the vagina and / or parameters) , radiotherapy associated with curietherapy , plays a major role. Until recently this association was the standard treatment for advanced stage uterine cancer. With this combination, rates of local failures (evolutionary prosecution and local recurrences) were 20 to 50% in stages IIb and 50-75 % for stage III. More than 50% for patients with a cervical cancer locally advanced (FIGO stages II / IV) . The standard treatment, external radiotherapy followed by curietherapy allows expect survival rates at 5 years for approximately 30-45 %. For ten years, numerous studies have evaluated the addition of concurrent chemotherapy to radiotherapy in cancer of the cervix. More than 19 randomized trials have been published. A meta-analysis of these trials was undertaken to assess the role of radiochemotherapy in cancers of the cervix. The first meta-analysis published by the Cochrane Collaborative Group, taking into account 4580 patient, shows an improvement in survival, both in terms of progression free survival and overall survival for patients treated with radio chemotherapy respectively 16% and 12 % (p < 0.0001). The rate of metastasis is also decreased (p < 0.0001). Survival rates were significantly better when platinum salt was used ( p < 0.0001 ) . However, no clinical benefit of chemoradiotherapy has been demonstrated for tumors stages [1, 2] locally advanced, possibly due to small number of patients. The investigators have previously shown that antiviral agents used in preclinical models, Cidofovir® causes the selective radiosensitization of cells infected by the papillomavirus (HPV). This trial proposes to study a new concept to increase radiochemotherapy efficiency: the modulation of the expression of viral oncoproteins HPV virus by an antiviral agent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cervix cancer : Squamous cell carcinoma or adenocarcinoma of stage IB2> 4 cm, II, III or IVA (International Federation of Gynecology Obstetrics, regardless of pelvic lymph node status (optional surgical exploration) without paraaortic metastasis.
2. Detection of the virus genome of HPV positive on the primary tumor.
3. General state ECOG performance status 0-1.
4. 18 </ = age </ = 70 years.
5. PN> 2000 / mm3
6. hemoglobin> 9 g/l after transfusion if necessary .
7. platelets > 100 000 / mm3
8. Serum creatinine <1.5 upper limit of normal.
9. Liver function tests (SGOT, SGPT, alkaline phosphatase and bilirubin) <1.5 upper limit of normal.
10. Life expectancy> 3 months.
11. Systematic Beta HCG Dosage for premenopausal women.
12. Informed consent signed after informing the patient.
13. Proteinuria <2g / L (200mg / dL) and creatinine clearance of> / = 55 ml / min.

Exclusion Criteria:

1. Other histological types of cervix tumor than those mentioned in the inclusion criteria.
2. Search of viral sequences on the negative HPV tumor diagnosis.
3. History of cancer other than basal cell carcinoma.
4. Pre-treatment with radiotherapy or chemotherapy.
5. Ongoing pregnancy.
6. History or active psychiatric illness.
7. Nephropathy whatever the grade.
8. Infection scalable.
9. Active infection or other serious underlying pathology may prevent the patient receiving the treatment (in particular hepatic or cardiac).
10. Inclusion in another clinical trial protocol with an experimental molecule (during the study or within one month before inclusion).
11. Inability to submit to medical monitoring study for geographical, social or psychological.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Assessed every week after inclusion up to 10 weeks

SECONDARY OUTCOMES:
Efficacy Using RECIST criteria | Assessed 14 weeks after inclusion
  Using RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France